CLINICAL TRIAL: NCT07390994
Title: Prognostic Impact of PHENOtyping de Novo Coronary Artery Disease Prior to Drug-Coated Balloon Angioplasty by Optical Coherence Tomography (PICCOLETO IX PHENO)
Brief Title: The PICCOLETO IX PHENO Study
Acronym: PIX-PHENO
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Ricerca e Innovazione Cardiovascolare ETS (Other)
Responsible Party: Sponsor
Other Study IDs: PICCOLETO IX - PHENO
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug-Coated Balloon; Optical Coherence Tomography; Percutaneous Coronary Intervention; Plaque phenotype
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate whether pre-procedural OCT-derived de novo coronary lesion phenotype (lipid-rich, fibrotic, calcific; and ACS mechanisms such as plaque rupture/erosion/calcified nodule) is associated with clinical outcomes after DCB angioplasty.

DETAILED DESCRIPTION:
PICCOLETO IX PHENO is an investigator-initiated, multicenter, international, ambispective (retrospective and prospective) cohort study enrolling patients who underwent DCB angioplasty for de novo coronary artery disease with preprocedural OCT assessment of the target segment. OCT images (baseline mandatory; post-preparation and post-PCI when available) and angiography will be analyzed by independent core laboratories; clinical events will be adjudicated by an independent committee. The primary endpoint is clinically-driven target lesion revascularization at 12 months; secondary endpoints include device-oriented composite endpoint (cardiac death, TLR, target-vessel MI), target vessel revascularization, MI endpoints, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary syndrome or acute coronary syndrome diagnosis (per ESC guidelines).
* De novo obstructive CAD: ≥50% left main stenosis, or any stenosis ≥70%, or FFR <0.80 in any other major epicardial vessel, or MLA deemed ischemic at intravascular imaging.
* OCT assessment of the target segment phenotype prior to lesion preparation and DCB angioplasty.
* Successful DCB angioplasty according to DCB ARC criteria.
* Patients who underwent DCB-only PCI, or hybrid DCB-DES PCI with at least 20 mm of the target segment treated with DCB.

Exclusion Criteria:

* Previous revascularization of the target segment with stent.
* Hybrid DCB-DES PCI with DCB-treated segment <20 mm and/or lacking complete OCT assessment of the DCB-treated segment and/or bailout stenting.
* Lack of at least 6 months of clinical follow up.
* PCI of chronic total occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic coronary syndrome or acute coronary syndrome who underwent drug-coated balloon angioplasty for de novo obstructive coronary artery disease with preprocedural optical coherence tomography assessment of the target segment.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
Clinically-driven Target Lesion Revascularization (TLR) | 12 months
  Any repeat revascularization (percutaneous or surgical) of the target lesion performed for recurrent symptoms or objective evidence of ischemia attributable to the target lesion.

SECONDARY OUTCOMES:
Device-Oriented Composite Endpoint (DOCE) | 12 months
  Composite of cardiac death, target-vessel myocardial infarction, and clinically-driven target lesion revascularization.
Target Vessel Revascularization (TVR) | 12 months
  Any repeat revascularization (percutaneous or surgical) of the target vessel.
All-cause Mortality | 12 months
  Death from any cause during the study follow-up period.
Cardiac Death | 12 months
  Death attributed to cardiovascular causes, including death from unknown cause.
Target-Vessel Myocardial Infarction (TV-MI) | 12 months
  Myocardial infarction attributable to the target vessel based on clinical, electrocardiographic, and biomarker criteria according to the Fourth Universal Definition of Myocardial Infarction.
Any Myocardial Infarction | 12 months
  Any myocardial infarction (target-vessel or non-target-vessel) according to the Fourth Universal Definition of Myocardial Infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Luca Gurgoglione, Principal Investigator — A.O.U. di Parma

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may be made available to qualified researchers upon reasonable request after study completion and primary publication, subject to appropriate data use agreements and ethics committee approval.